CLINICAL TRIAL: NCT05500924
Title: The Effects of Ankle Mulligan Mobilization on Range of Motion, Balance, Functional Performance and Quality of Life of Children With Diplegic Spastic Cerebral Palsy
Brief Title: Effects of Ankle Mobilization on Body Structure, Function, Activities and Participation of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2022-0160
Record Dates: First submitted 2022-08-04; First posted 2022-08-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Diplegic Cerebral Palsy With Spasticity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 5 sets of functional activities each will be repeated for 3 times , while the therapist is performing mulligan mobilization techniques Sit to stand Squat Stand to sit Stairs stepping Bridging
  Interventions: Other: Intervention group
- Control group (Experimental): 5 sets of functional activities each will be repeated for 3 times: Sit to stand Squat Stand to sit Stairs stepping Bridging
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — 5 sets of functional activities each will be repeated for 3 times , while the therapist is performing mulligan mobilization techniques Sit to stand Squat Stand to sit Stairs stepping Bridging

SUMMARY:
Cerebral palsy is the most common motor disability of childhood (Suvanand et al 1997). By definition CP is a static encephalopathy, but the musculoskeletal pathology is a major concern . Chronic neurologic impairment affects the development of bones and muscles. In spastic hemiplegia, the affected side demonstrates muscle atrophy and limb shortening, compared to the unaffected side. Thus, CP is a neuromusculoskeletal disorder . Musculoskeletal conditions of people with CP can develop or worsen across the lifespan as a consequence of the primary neuromotor impairments which will affect their physical activity and participation. In fact these complications can lead to lose the ability of walking in ambulatory children up to 30% . (Peterson 2015) Physical inactivity among regularly growing paediatric community has become a general health load.

Neurological interventions are well documented, However, there is a gap of information and evidence documenting the orthopaedic intervention effect on orthopaedic secondary complications in CP. Even though the neurological pathology isn't progressive , the orthopaedic complication itself is progressive and affect the ability of the CP children to progress, and in so many cases they lose their functional achievements when their functional status can't meet their growth requirements any more, due to the neurological dysfunction and progressive secondary complications, that makes walking less efficient , less effective, and increased fatigue levels in gait. (Tosi et al. 2009).

Little is known about the practice of Brian Mulligan's mobilization with movement (MWM) in CP patients in early ages, for the secondary complication of the ankle hypomobility and ROM. This study will be conducted to discover the immediate effect of MWM on the ankle to improve the range and mobility of ankle as a musculoskeletal (dysfunction) for the function of gait.

DETAILED DESCRIPTION:
Cerebral palsy is the most common motor disability of childhood (Suvanand et al 1997). By definition CP is a static encephalopathy, but the musculoskeletal pathology is a major concern . Chronic neurologic impairment affects the development of bones and muscles. In spastic hemiplegia, the affected side demonstrates muscle atrophy and limb shortening, compared to the unaffected side. Thus, CP is a neuromusculoskeletal disorder . Musculoskeletal conditions of people with CP can develop or worsen across the lifespan as a consequence of the primary neuromotor impairments which will affect their physical activity and participation. In fact these complications can lead to lose the ability of walking in ambulatory children up to 30% . (Peterson 2015) Physical inactivity among regularly growing paediatric community has become a general health load.

Neurological interventions are well documented, However, there is a gap of information and evidence documenting the orthopaedic intervention effect on orthopaedic secondary complications in CP. Even though the neurological pathology isn't progressive , the orthopaedic complication itself is progressive and affect the ability of the CP children to progress, and in so many cases they lose their functional achievements when their functional status can't meet their growth requirements any more, due to the neurological dysfunction and progressive secondary complications, that makes walking less efficient , less effective, and increased fatigue levels in gait. (Tosi et al. 2009).

Little is known about the practice of Brian Mulligan's mobilization with movement (MWM) in CP patients in early ages, for the secondary complication of the ankle hypomobility and ROM. This study will be conducted to discover the immediate effect of MWM on the ankle to improve the range and mobility of ankle as a musculoskeletal (dysfunction) for the function of gait.

Research questions What is the effect of Ankle MWM in functional activities on gait function ? What is the effect of Ankle MWM in functional activities on balance function ? What is the effect of Ankle MWM in functional activities on quality of life? What is the effect of Ankle MWM in functional activities on fatigue?

Research hypothesis Ankle MWM in functional activities improves gait function? Ankle MWM in functional activities improve balance? Ankle MWM in functional activities improves quality of life? Ankle MWM in functional activities increase happiness? Research objectives To investigate the effect of Ankle MWM in functional activities on gait function? To study the effect of Ankle MWM in functional activities on balance function? To highlight the effect of Ankle MWM in functional activities on quality of life? To study the effect of Ankle MWM in functional activities on happiness?

ELIGIBILITY:
Inclusion Criteria:

* Spastic Diplegic CP
* healthy bones appropriate for mobilisation
* ages between 4-14
* GMFCS I, II
* Ashworth scale 2-3 (For Gastrocnemius Muscle)
* Good cognitive ability to understand the orders in the tests
* CP children who continued to take regular physiotherapy sessions

Exclusion Criteria:

* Recent correcting orthopaedic surgeries until 6 months before recruitment
* Children received or intending to receive Botox within an interval of 3 months
* Children who have full Ankle dorsal flexion.
* fixed contracture

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Change of Ankle Range of Motion | Baseline and post 4 weeks assessment
  ROM of Ankle Dorsiflexion passively and actively will be done using goniometer to assess any changes.
Change in the Six minutes walking test: The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface | Baseline and post 4 weeks assessment
  For measuring the changes in walking activities.The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
Change inTime up and go (TUG) test: The TUG test is a reliable and responsive measure of balance and mobility for children with CP | Baseline and post 4 weeks assessment
  For assessing the change in Balance and mobility
Change in the Pediatric Quality of Life: it is measured by measure by CP-specific questionnaire. We will use The Arabic-CP-QOL-questionnaire | Baseline and post 4 weeks assessment
  To assess the change in the quality of life and happiness of the children
Change in the Gross Motor Function Measure (GMFM) scale which is designed to measure changes in gross motor function over time or with intervention in children with cerebral palsy. | Baseline and post 4 weeks assessment
  To assess the changes in the Functional performance in thegross motor function of Cerebral Palsy children

CONTACTS AND LOCATIONS:
Overall Officials: Zehra G. Topco, PhD, Study Director — Eastern Medeterranean University
Locations (1):
- Palestine Ahliya university, Bethlehem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ragheb Abushameh RS, Topcu ZG, Tunal AN, Amro A, Arab AA. The effects of ankle mulligan mobilisation in children with cerebral palsy: A randomized single blind control study. J Pak Med Assoc. 2024 Jul;74(7):1219-1223. doi: 10.47391/JPMA.10328. PMID 39028043